CLINICAL TRIAL: NCT05689034
Title: A Multicenter Randomized Double-blind Placebo-controlled Study to Investigate Azvudine in Symptomatic Adult Participants With COVID-19 Who Are at Increased Risk of Progressing to Severe Illness
Brief Title: Multicenter Randomized Double-blind Placebo-controlled Study to Investigate Azvudine in Symptomatic Adults With COVID-19 at Increased Risk of Progressing to Severe Illness
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FNC-K3482
Record Dates: First submitted 2023-01-17; First posted 2023-01-18 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-08

CONDITIONS: COVID-19 Respiratory Infection
MeSH Terms: interventions — azvudine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized, Double-blind, Placebo-controlled Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azvudine (Active Comparator): Azvudine in Patients at Potential Risk of Progressing to Severe COVID-19 Infection
  Interventions: Drug: Azvudine
- Placebo (Placebo Comparator): Placebo in Patients at Potential Risk of Progressing to Severe COVID-19 Infection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azvudine — Azvudine po. 5mg daily for 7 days
  Arms: Azvudine
Drug: Placebo — Placebo po. 5 tablets daily for 7 days
  Arms: Placebo

SUMMARY:
To investigate whether treatment with Azvudine reduces the risk of severe illness or death in patients who are at a potential risk of progressing to severe COVID-19 infection.

DETAILED DESCRIPTION:
The study is designed as a randomized, parallel, double-blind, placebo-controlled trial, in which all participants will be randomized to a test group or control group in a 1:1 ratio.

The test group will be given Azvudine in combination with conventional therapy excluding anti-viral therapy and observed for efficacy. The control group will be given placebo in combination with conventional therapy excluding anti-viral therapy and observed for efficacy.

Test Group will recruit 548 participants who will be given Azvudine + conventional therapy other than antiviral*5 mg/day, oral, up to 7 days (1 mg/tablet).

Control Group will recruit 548 who will be given Placebo + conventional therapy other than antiviral* 5 tablets/day, oral, up to 7 days.

ELIGIBILITY:
Inclusion Criteria:

* (1) An age of 18 years or over (inclusive); (2) Not more than five days since the development of COVID-19 symptoms, and positive for nucleic acid or antigen test for COVID-19 within five days before enrollment; (3) Presence of at least one symptom related to COVID-19 infection at the time of enrollment; (4) Agreement to practice effective birth control (for females of child-bearing potential); (5) Presence of at least one high risk factor for severe COVID-19 infection:

  * Age ≥ 60 years;

    * BMI>25；

      * Fever (body temperature ≥ 38℃) for ≥ 3 days;

        * Current smokers (still being smoking within 30 days before enrollment and have used at least 100 cigarettes up to date);

          * Immunosuppressive diseases, including but not limited to: myelosuppression or organ transplantation or primary immunodeficiency disease; prolonged use of immunosuppressive agents (≥ 20 mg/d for at least 14 days in the case of prednisone within the last 30 days); biologic therapy (such as infliximab, etc.); use of immunomodulators (including but not limited to methotrexate, azathioprine, etc.); radiotherapy and/or chemotherapy for any malignancies within 90 days (for chest radiotherapy, this time interval should be more than 6 months);

            * Chronic lung disease (such as asthma requiring intervention daily, bronchiectasis, COPD, pulmonary hypertension, OSAS, interstitial lung disease, etc.);

              * Hypertension; ⑧ Cardiovascular diseases (previously diagnosed as myocardial infarction or stroke, TIA (transient ischemic attack), cardiac insufficiency, angina pectoris requiring nitrate therapy, CABG, post-PCI, post-carotid endarterectomy and aortic bypass surgery, etc.);

                ⑨ Type 1 or type 2 diabetes;

                ⑩ Neurodevelopmental abnormalities (such as cerebral palsy, Down's syndrome) or other genetic or metabolic syndromes and severe congenital malformations;

                ⑪ Active tumors (excluding localized skin cancer);

                ⑫ No vaccination against COVID-19

Exclusion Criteria:

* (1) Known or suspected allergy to the components of Azvudine Tablets; (2) Patients diagnosed as severe or critical COVID-19 infection (Severe: 1. shortness of breath with RR ≥ 30 breaths/min; 2. oxygen saturation ≤ 93% when inhaling air at rest; 3. partial pressure of arterial oxygen (PaO2) / fraction of inspired oxygen (FiO2) ≤ 300 mmHg; 4. progressive worsening of clinical symptoms, and obvious lesion progression > 50% on lung images within 24 to 48 hours. Critical: 1. respiratory failure, requiring mechanical ventilation; 2. shock; 3. concomitant organ failure, requiring care in ICU); (3) Patients with severe liver disease (total bilirubin [TBIL] ≥ 2 × upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 3 × ULN; (4) Patients with severe renal insufficiency (glomerular filtration rate ≤ 60 mL/min/1.73 m2) or currently on continuous renal replacement therapy, hemodialysis, and/or peritoneal dialysis; (5) Patients with malabsorption syndrome or any other condition compromising gastrointestinal absorption, or patients requiring parenteral nutrition or with difficulty in taking the investigational product orally; (6) Known HIV infection; (7) Presence of diabetic ketosis or hyperosmolar hyperglycemic state (HHS); (8) Total neutrophil count < 750 cells/L; (9) Pregnant or lactating women or those who plan to have a child during participation in this study and within six months after the end of this study; (10) Currently participating in another clinical trial or currently using another investigational product; (11) Presence of other active infections (must be etiologically confirmed) in addition to COVID-19 infection; (12) Presence of any comorbidities requiring hospitalization and/or a surgical procedure within 7 days prior to the start of this study or a comorbidity considered life-threatening within 30 days prior to the start of this study; (13) Patients who have received or are expected to receive convalescent plasma for COVID-19; (14) Previous treatment with anti-viral agents that have been proved to be effective against COVID-19, including but not limited to Nirmatrelvir/Ritonavir or Molnupiravir (this criterion does not apply to use of glucocorticoids for reasons other than COVID-19); (15) Other conditions that make it inappropriate for the participant to take part in this trial at the investigator's discretion.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1096 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of COVID-19-related critical illness or all-cause death within 28 days. | 28 days
  Proportion of COVID-19-related critical illness or all-cause death within 28 days.
  COVID-19-related critical illness is defined as: a patient with an SpO2 of 90% to 95% requiring high-flow oxygen inhalation with a fraction of inspired oxygen (FiO2) not less than 60% or requiring non-invasive ventilation with a FiO2 not less than 60%; or requiring mechanical ventilation or ECMO for organ support.

SECONDARY OUTCOMES:
Incidence rates of Azvudine-related adverse events and serious adverse events | 28 days
  Incidence rates of Azvudine-related adverse events and serious adverse events
Duration of COVID-19-related symptoms | 14 days
  Duration of COVID-19-related symptoms
All-cause death | 6 months
  All-cause death
COVID-19 viral load in pharyngeal swabs | D1, D3, D7
  COVID-19 viral load in pharyngeal swabs
Days of hospitalization and ICU stay | 28 days
  Days of hospitalization and ICU stay

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory and Critical Care Medicine, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tian X, Xu Y, Wang L, Dong C, Yan X, Fan J, Xie H, Zhang H, Wang J, Liu Y, Wang Y, Pan S, Wu A, Liu X, Yao C, Wang M. Efficacy and safety of azvudine in symptomatic adult COVID-19 participants who are at increased risk of progressing to critical illness: a study protocol for a multicentre randomized double-blind placebo-controlled phase III trial. Trials. 2024 Jan 22;25(1):77. doi: 10.1186/s13063-024-07914-3. PMID 38254211